CLINICAL TRIAL: NCT00016718
Title: An Open-Label Study to Evaluate the Safety, Tolerance, Antiviral Activity, and Pharmacokinetics of Emtricitabine in Combination With Efavirenz and Didanosine in a Once-Daily Regimen in HIV Infected, Antiretroviral Therapy Naive or Very Limited Antiretroviral Exposed Pediatric Subjects
Brief Title: Safety and Effectiveness of Emtricitabine, Efavirenz, and Didanosine in HIV Infected Children Who Have Taken Few or No Anti-HIV Drugs
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P1021; 10038 (Registry Identifier: DAIDS ES); ACTG P1021; PACTG P1021; IMPAACT P1021
Record Dates: First submitted 2001-05-31; First posted 2001-08-31 (Estimated); Results first posted 2017-10-17 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2017-09

CONDITIONS: HIV Infections
Keywords: Didanosine; Drug Therapy, Combination; Drug Administration Schedule; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Pharmacokinetics; Deoxycytidine; Efavirenz; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — Didanosine; efavirenz; Emtricitabine; Racivir

STUDY DESIGN:
Masking Description: open-label

ARMS (3):
- Age Group 1: 90 days to < 3 years of age (FTC, EFV, ddI) (Experimental): Emtricitabine (FTC), Efavirenz (EFV) and Didanosine (ddI) together once daily
  Interventions: Drug: Didanosine (ddI); Drug: Efavirenz (EFV); Drug: Emtricitabine (FTC)
- Age Group 2: 3 to 12 years of age (FTC, EFV, ddI) (Experimental): Emtricitabine (FTC), Efavirenz (EFV) and Didanosine (ddI) together once daily
  Interventions: Drug: Didanosine (ddI); Drug: Efavirenz (EFV); Drug: Emtricitabine (FTC)
- Age Group 2: 13 to 21 years of age (FTC, EFV, ddI) (Experimental): Emtricitabine (FTC), Efavirenz (EFV) and Didanosine (ddI) together once daily
  Interventions: Drug: Didanosine (ddI); Drug: Efavirenz (EFV); Drug: Emtricitabine (FTC)

INTERVENTIONS:
Drug: Didanosine (ddI) — Antiretroviral Didanosine (ddI) : 240 mg/m^2 up to a maximum of 400 mg once daily
  Other Names: Videx, Videx EC
Drug: Efavirenz (EFV) — Antiretroviral For Age Group 1 Efavirenz (EFV): dose adjusted for body size and for Age Groups 2 and 3 Efavirenz (EFV): up to a maximum of 600 mg once daily as a capsule ot 720 mg as an oral solution
  Other Names: Sustiva
Drug: Emtricitabine (FTC) — Antiretroviral Emtricitabine (FTC): 6 mg/Kg up to a maximum of 200 mg once daily
  Other Names: Emtriva

SUMMARY:
Treatment of HIV-infected patients involves combining drugs from different classes of anti-HIV drugs. One preferred regimen for adults is 2 nucleoside reverse transcriptase inhibitors (NRTIs) and 1 protease inhibitor (PI). For children, this regimen may be too complicated or the drugs may be too difficult to take by mouth. The purpose of this study was to determine the long-term safety and effectiveness of daily didanosine (ddI), efavirenz (EFV), and emtricitabine (FTC) in pediatric patients who had taken few or no anti-HIV drugs.

DETAILED DESCRIPTION:
Anti-HIV treatment options are limited for pediatric patients because combination therapies recommended for adults may not be appropriate for children or adolescents. Few PIs are available in formulations appropriate for pediatric patients, and complex dosing schedules and food requirements may be detrimental to treatment adherence. A once-daily regimen of the NRTIs ddI and FTC and the nonnucleoside reverse transcriptase inhibitor (NNRTI) EFV has been shown safe and well tolerated in adults.

This Phase I/II open label study evaluated the long-term safety and efficacy of a ddI, FTC, and EFV regimen in pediatric patients. All study patients were either absolutely naive to antiretroviral therapy or had received less than or equal to 56 days perinatal prophylaxis or less than 7 days of cumulative antiretroviral therapy prior to study entry, and had a plasma screening plasma HIV-1 RNA levels >= 5000 copies/mL. This study was written to characterize the disposition of FTC, determine the PK data for ddI-EC QD, comparing the bio-availability of the enteric coated formulation with ddI pediatric powder for oral solution, and to provide insight into the age related pharmacokinetics differences observed in this and other studies.

HIV infected pediatric patients were stratified into three age Groups: Group 1: 90 days to <3 years of age; Group 2: 3 years to 12 years of age (inclusive); and Group 3: 13 to 21 years of age (inclusive). The initial study doses for the triple drug regimen was FTC, 6 mk/kg up to a maximum of 200 mg once daily, for EFV, the dose for age Group 1 was determined in PACTG 382 and dose adjusted for body size, and the doses for age Groups 2 and 3 were defined in the dosing table of the protocol of up to a maximum of 600 mg once daily as a capsule or 720 mg as an oral solution; for ddI, 240 mg/m2 up to a maximum of 400 mg once daily. Comparison of age groups was not required as per the protocol.

Patients were followed for a maximum of 192 weeks; all patients were to receive ddI, EFV, and FTC together once daily. Study visits occurred at study entry, Weeks 2,and 4, and every 4 weeks thereafter. Blood collection, medical history assessment, and a physical exam occurred at all visits; urine collection occurred at selected visits. Intensive pharmacokinetic (PK) studies was done at Weeks 2 and 12 to determine if dose adjustments were required for any of the drugs. If virologic failure was determined, PK studies was repeated 4 weeks after adjustments in therapy. Parents or guardians were asked to complete treatment adherence questionnaires at some visits. Some patients were also asked to participate in an additional PK study after Week 16 or week 96.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* Antiretroviral naive OR have received no more than 56 days of drugs to prevent mother-to-child transmission of HIV OR have received less than 7 total days of antiretroviral therapy
* Viral load of 5,000 copies/ml or more
* Any Center for Disease Control (CDC) classification and immune status
* Able to swallow study medications
* Parent or guardian willing to provide informed consent, if applicable
* Willing to use acceptable forms of contraception
* female subjects of childbearing potential with a negative serum beta human chronic gonadotropin

Exclusion Criteria:

* Allergic to study medications or their formulations
* Kidney disease
* Positive for hepatitis B or C
* Acute opportunistic infection (OI) or bacterial infection requiring treatment at study entry
* Taking drugs to treat tuberculosis
* Taking anti-HIV drugs other than those included in this study
* Hemoglobin >= grade 3 at screening
* Absolute Neutrophil counts >= grade 2 at screening
* Platelets >= Grade 2 at screening
* Bilirubin >= Grade 2 at screening
* SGOT (AST), SGPT(ALT) >= Grade 2 at screening
* Non-fasting triglycerides >= Grade 2 at screening. Confirmed by a 2nd determination >=100 mg/dl at fasting state
* Pancreatic amylase or total amylase+ lipase >= Grade 2 at screening
* Taking any investigational drugs
* Anti-cancer drugs within 1 year of study screening
* Serious medical event within 21 days of study screening
* Active or history of pancreatitis
* Require certain medications. Patients requiring short courses of steroids (less than 14 days) for asthma are not excluded.
* Active or history of significant peripheral neuropathy
* Difficulty with food or severe chronic diarrhea within 30 days before study entry
* Unable to eat at least 1 meal per day (or to feed at least 3 times per day, for infants) because of chronic nausea, vomiting, swallowing problems, or stomach upset
* Unable to swallow oral medications
* Pregnant or breastfeeding

Ages: 90 Days to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 2001-08; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ross E. McKinney, Jr., MD, Study Chair — Duke University; Mobeen H. Rathore, MD, Study Chair — Pediatric Infectious Diseases/Immunology, University of Florida Health Science Center
Locations (18):
- United States (16):
  - UCSD Maternal, Child, and Adolescent HIV CRS, San Diego, California
  - UCSF Pediatric AIDS CRS, San Francisco, California
  - Univ. of Colorado Denver NICHD CRS, Aurora, Colorado
  - Howard Univ. Washington DC NICHD CRS, Washington D.C., District of Columbia
  - Univ. of Florida Jacksonville NICHD CRS, Jacksonville, Florida
  - Univ. of Miami Ped. Perinatal HIV/AIDS CRS, Miami, Florida
  - Chicago Children's CRS, Chicago, Illinois
  - Rush Univ. Cook County Hosp. Chicago NICHD CRS, Chicago, Illinois
  - Children's Hosp. of Boston NICHD CRS, Boston, Massachusetts
  - WNE Maternal Pediatric Adolescent AIDS CRS, Worcester, Massachusetts
  - Nyu Ny Nichd Crs, New York, New York
  - Harlem Hosp. Ctr. NY NICHD CRS, New York, New York
  - SUNY Upstate Med. Univ., Dept. of Peds., Syracuse, New York
  - DUMC Ped. CRS, Durham, North Carolina
  - St. Jude/UTHSC CRS, Memphis, Tennessee
  - Texas Children's Hosp. CRS, Houston, Texas
- Puerto Rico (2):
  - Univ. of Puerto Rico Ped. HIV/AIDS Research Program CRS, San Juan
  - San Juan City Hosp. PR NICHD CRS, San Juan

REFERENCES:
- [Background] McKinney RE Jr, Cunningham CK. Newer treatments for HIV in children. Curr Opin Pediatr. 2004 Feb;16(1):76-9. doi: 10.1097/00008480-200402000-00014. PMID 14758118
- [Result] Weinberg A, Dickover R, Britto P, Hu C, Patterson-Bartlett J, Kraimer J, Gutzman H, Shearer WT, Rathore M, McKinney R; PACTG 1021 team. Continuous improvement in the immune system of HIV-infected children on prolonged antiretroviral therapy. AIDS. 2008 Nov 12;22(17):2267-77. doi: 10.1097/QAD.0b013e3283189bb3. PMID 18981766

RESULTS

PARTICIPANT FLOW:
Groups:
- Age Group 1: 90 days to < 3 years of age, inclusive (FTC, EFV, ddI)
- Age Group 2: 3 years to 12 years of age, inclusive (FTC, EFV, ddI)
- Age Group 3: 13 years to 21 years of age, inclusive (FTC, EFV, ddI)
Period: Overall Study
Arm/Group | Age Group 1 | Age Group 2 | Age Group 3
Started | 6 | 21 | 16
Completed | 6 | 21 | 16
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Age Group 1 | Age Group 2 | Age Group 3 | Total
Number analyzed (Participants) | 6 | 21 | 16 | 43
Age, Continuous [Median (Full Range); unit: years] | 0.5 [0.3 to 2.6] | 5.7 [3.2 to 11.7] | 17.5 [14.5 to 21.1] | 9.6 [0.3 to 21.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 11 | 6 | 21
  Male | 2 | 10 | 10 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White non-Hispanic | 0 | 3 | 2 | 5
  Black non-Hispanic | 4 | 11 | 12 | 27
  Hispanic | 2 | 7 | 2 | 11

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Who Developed Grade 3 or 4 Adverse Events Attributed to the Study Treatment.
Description: Adverse events were graded using the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 1.0, December 2004, Clarification August 2009, which is available on the RCC website at (http://rcc.tech-res.com/). Adverse Events of Grade 3 or 4 laboratory abnormalities or signs and symptoms that were judged by the study team to be possibly or probably related to the study treatment.
  Comparisons between age groups were not required as per protocol.
Time Frame: At study entry, weeks 2 and 4, every 4 weeks up to week 96 and every 6 weeks thereafter for Group 1 participants and at study entry, weeks 2 and 4, every 4 weeks up to week 144 and every 12 weeks thereafter for Groups 2 and 3
Population: All Participant who enrolled in the study
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Age Group 1 | Age Group 2 | Age Group 3
Number analyzed (Participants) | 6 | 21 | 16
proportion of participants | 0.17 [0.03 to 0.56] | 0.1 [0.03 to 0.29] | 0.19 [0.07 to 0.43]

2. Primary Outcome: Proportion of Participants With Suppression of HIV Viral Load to Less Than 400 Copies/ml at Week 16
Description: Proportion was calculated as number of participants with HIV-1 RNA <= 400 copies/ml relative to the number of participants with HIV-1 RNA measured at that time point.
Time Frame: At week 16
Population: All Participant who enrolled in the study and with available HIV-RNA at week 16
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Age Group 1 | Age Group 2 | Age Group 3
Number analyzed (Participants) | 6 | 21 | 16
proportion of participants | 0.83 [0.36 to 0.99] | 0.86 [0.64 to 0.97] | 0.81 [0.54 to 0.96]

3. Primary Outcome: Proportion of Participants With Suppression of HIV Viral Load to Less Than 50 Copies/ml at Week 16
Description: Proportion was calculated as number of participants with HIV-1 RNA <= 50 copies/ml relative to the number of participants with HIV-1 RNA measured at that time point.
Time Frame: At week 16
Population: All Participant who enrolled in the study and with available HIV-RNA at week 16
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Age Group 1 | Age Group 2 | Age Group 3
Number analyzed (Participants) | 6 | 21 | 16
proportion of participants | 0.50 [0.12 to 0.88] | 0.76 [0.53 to 0.92] | 0.75 [0.48 to 0.93]

ADVERSE EVENTS:
Time Frame: At study entry, weeks 2 and 4, every 4 weeks up to week 96 and every 6 weeks thereafter for Group 1 participants and at study entry, weeks 2 and 4, every 4 weeks up to week 144 and every 12 weeks thereafter for Group 2 and 3 participants
Description: The study protocol required reporting of all new diagnoses, signs/symptoms and laboratory events .Adverse events were graded using the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 1.0, December 2004, Clarification August 2009, which is available on the RCC website at (http://rcc.tech-res.com/).
Groups:
- Age Group 1: 90 days to 3 years of age, inclusive (FTC, EFV, ddI)
Arm/Group | Age Group 1 | Age Group 2 | Age Group 3
Serious Adverse Events (participants affected / at risk) | 1/6 | 4/21 | 5/16
Other Adverse Events (participants affected / at risk) | 6/6 | 21/21 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Age Group 1 (N=6) | Age Group 2 (N=21) | Age Group 3 (N=16)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 2
Blood glucose decreased (Investigations) | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0
Liver function test increased (Investigations) | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Age Group 1 (N=6) | Age Group 2 (N=21) | Age Group 3 (N=16)
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 4
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Cerebral palsy (Congenital, familial and genetic disorders) | 1 | 0 | 0
Congenital nystagmus (Congenital, familial and genetic disorders) | 1 | 0 | 0
Microcephaly (Congenital, familial and genetic disorders) | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 3 | 1
Otorrhoea (Ear and labyrinth disorders) | 1 | 1 | 0
Tympanic membrane hyperaemia (Ear and labyrinth disorders) | 1 | 1 | 0
Blepharospasm (Eye disorders) | 0 | 0 | 1
Blindness (Eye disorders) | 1 | 0 | 0
Eye discharge (Eye disorders) | 2 | 1 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0 | 0
Pupil fixed (Eye disorders) | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 5 | 4 | 0
Gastritis (Gastrointestinal disorders) | 0 | 2 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 2
Gingival hypertrophy (Gastrointestinal disorders) | 1 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 4
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 2
Vomiting (Gastrointestinal disorders) | 3 | 1 | 3
Asthenia (General disorders) | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 1
Dysplasia (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1
Localised oedema (General disorders) | 0 | 0 | 1
Mass (General disorders) | 0 | 0 | 1
Peripheral swelling (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 3 | 7 | 3
Secretion discharge (General disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Acarodermatitis (Infections and infestations) | 0 | 4 | 1
Acute sinusitis (Infections and infestations) | 0 | 4 | 7
Atypical mycobacterial lymphadenitis (Infections and infestations) | 0 | 0 | 1
Bacterial vaginosis (Infections and infestations) | 0 | 0 | 1
Body tinea (Infections and infestations) | 0 | 3 | 4
Bronchitis (Infections and infestations) | 1 | 0 | 2
Cellulitis (Infections and infestations) | 0 | 1 | 1
Cervicitis human papilloma virus (Infections and infestations) | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 2 | 0 | 0
Coxsackie viral infection (Infections and infestations) | 1 | 0 | 0
Epididymitis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 5 | 1
Gastroenteritis rotavirus (Infections and infestations) | 1 | 0 | 0
Genital herpes simplex (Infections and infestations) | 0 | 0 | 1
Genital infection bacterial (Infections and infestations) | 0 | 0 | 1
Gingivitis (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 1
Impetigo (Infections and infestations) | 0 | 5 | 0
Latent tuberculosis (Infections and infestations) | 0 | 0 | 1
Onychomycosis (Infections and infestations) | 0 | 0 | 2
Oral candidiasis (Infections and infestations) | 0 | 2 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 1
Otitis externa (Infections and infestations) | 0 | 2 | 0
Otitis media (Infections and infestations) | 1 | 8 | 0
Otitis media acute (Infections and infestations) | 1 | 5 | 0
Otitis media bacterial (Infections and infestations) | 1 | 0 | 0
Papilloma viral infection (Infections and infestations) | 0 | 0 | 1
Parotitis (Infections and infestations) | 0 | 2 | 0
Pharyngitis (Infections and infestations) | 0 | 3 | 1
Pneumonia (Infections and infestations) | 0 | 2 | 0
Purulent discharge (Infections and infestations) | 0 | 2 | 0
Salpingitis (Infections and infestations) | 0 | 0 | 1
Skin candida (Infections and infestations) | 1 | 0 | 0
Tinea capitis (Infections and infestations) | 1 | 4 | 0
Tinea cruris (Infections and infestations) | 0 | 0 | 1
Tinea infection (Infections and infestations) | 0 | 2 | 1
Tinea pedis (Infections and infestations) | 0 | 0 | 2
Trichomoniasis (Infections and infestations) | 0 | 0 | 1
Urethritis (Infections and infestations) | 0 | 0 | 1
Urethritis gonococcal (Infections and infestations) | 0 | 0 | 1
Urinary tract infection staphylococcal (Infections and infestations) | 0 | 0 | 1
Varicella (Infections and infestations) | 0 | 2 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 1
Vulvovaginitis (Infections and infestations) | 0 | 1 | 2
Vulvovaginitis trichomonal (Infections and infestations) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 3 | 12 | 5
Aldolase abnormal (Investigations) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 3 | 15 | 10
Blood alkaline phosphatase increased (Investigations) | 5 | 11 | 4
Blood bilirubin increased (Investigations) | 0 | 2 | 1
Blood calcium decreased (Investigations) | 0 | 9 | 1
Blood calcium increased (Investigations) | 4 | 0 | 3
Blood cholesterol increased (Investigations) | 4 | 16 | 11
Blood creatine phosphokinase abnormal (Investigations) | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 5 | 3
Blood creatinine increased (Investigations) | 0 | 10 | 12
Blood glucose abnormal (Investigations) | 0 | 1 | 1
Blood glucose decreased (Investigations) | 4 | 11 | 6
Blood glucose increased (Investigations) | 3 | 8 | 12
Blood magnesium decreased (Investigations) | 0 | 3 | 0
Blood potassium decreased (Investigations) | 0 | 6 | 9
Blood potassium increased (Investigations) | 5 | 8 | 4
Blood sodium decreased (Investigations) | 5 | 17 | 6
Blood sodium increased (Investigations) | 0 | 1 | 5
Blood triglycerides abnormal (Investigations) | 0 | 2 | 4
Blood triglycerides increased (Investigations) | 6 | 19 | 13
Blood urea abnormal (Investigations) | 0 | 5 | 1
Blood uric acid increased (Investigations) | 0 | 0 | 3
Haemoglobin decreased (Investigations) | 4 | 13 | 2
Neutrophil count decreased (Investigations) | 4 | 16 | 5
Pancreatic enzymes abnormal (Investigations) | 1 | 3 | 1
Total cholesterol/HDL ratio abnormal (Investigations) | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Coordination abnormal (Nervous system disorders) | 0 | 0 | 2
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Febrile convulsion (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 5
Hypertonia (Nervous system disorders) | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 2
Hypotonia (Nervous system disorders) | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1
Muscle spasticity (Nervous system disorders) | 1 | 0 | 0
Neurological symptom (Nervous system disorders) | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 2
Poor sucking reflex (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 2 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 2
Syncope (Nervous system disorders) | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 2
Bulimia nervosa (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 3
Insomnia (Psychiatric disorders) | 0 | 0 | 3
Major depression (Psychiatric disorders) | 0 | 0 | 1
Nightmare (Psychiatric disorders) | 0 | 3 | 2
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1 | 3
Polyuria (Renal and urinary disorders) | 0 | 0 | 1
Amenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 0 | 2
Genital lesion (Reproductive system and breast disorders) | 0 | 0 | 1
Penile discharge (Reproductive system and breast disorders) | 0 | 0 | 1
Scrotal pain (Reproductive system and breast disorders) | 0 | 0 | 1
Scrotal swelling (Reproductive system and breast disorders) | 0 | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1 | 2
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 8 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 4
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 2 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 2 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 2 | 4
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Scab (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 4 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.